CLINICAL TRIAL: NCT05859035
Title: Informational App Development for mHealth for Patient Self-Management of Opioid Use Disorder
Acronym: KIOS-I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biomedical Development Corporation (Industry)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-0232H; R42DA054881 (NIH)
Record Dates: First submitted 2023-04-13; First posted 2023-05-15 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KIOS Informational App evaluation (Experimental): Study participants will use the app at least three times per week. The app will contain a user interface that includes a login page, true/false questions for the user to answer, verified public domain educational information about drug and alcohol use, Likert-type questions regarding the information presented, and a closing "Thank You" screen.
  Interventions: Device: KIOS Informational App

INTERVENTIONS:
Device: KIOS Informational App — The KIOS informational app will contain a user interface that includes a login page, true/false questions for the user to answer, verified public domain educational information about drug and alcohol use, Likert-type questions regarding the information presented, and a closing "Thank You" screen.
  Other Names: KIOS-I

SUMMARY:
This study will evaluate the feasibility of an app that provides drug information to people in recovery from opioid use disorder. This study is designed to test the prototype app, not to determine health outcomes. The study will confirm the design and operating specifications prior to being evaluated in a larger clinical trial.

DETAILED DESCRIPTION:
The overall study is designed in two steps: 1) a one-week proof-of-concept study; and 2) a one-month pilot study.

Step 1: A one-week proof-of-concept study will be performed in a small population (n=5) of individuals in opioid use disorder recovery as an indicator of the app's suitability. Study participants will use the sham app for one week and will then complete a usability and user satisfaction survey. If the app is found to be exhibit acceptable usability and satisfaction, a one month study will be completed in a larger sample (see Step 2, below). If not, modifications to the app will be made and the one-week study will be repeated in a new group of participants.

Step 2: After completion of the proof-of-concept study, 20 new participants will be enrolled in a 4-week trial. Study participants will complete baseline assessments and then be asked to use the app at least three times per week, for four weeks. At the end of four weeks, participants will complete usability and user satisfaction surveys.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients 18 years of age or older
* Currently enrolled in an opioid treatment program and receiving medication assisted treatment for opioid use disorder
* Currently stable in opioid use disorder outpatient treatment for 4 weeks or longer
* Ability to access the app via smart phone, or tablet.

Exclusion Criteria:

* Unwilling or unable to comply with study requirements
* Have a psychiatric or medical disorder interfering with ability to use the app
* Incarcerated
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2024-01-10 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
Usability Score | The Systems Usability Scale will be administered at the end of one-week for participants enrolled in Step 1 of the study and at the end of four-weeks for participants enrolled in Step 2.
  The Systems Usability Scale-Modified is a non-health outcome, single-factor, 10-item self-report scale commonly used to evaluate participants' subjective experience using software. Systems Usability Scale yields a single number representing a composite measure of the overall usability of the system being studied. Systems Usability Scale scores have a range of 0 to 100, with higher scores representing a better outcome. Systems in early development may expect to have a rating of 30, while more mature systems should rate between 60 - 80.

SECONDARY OUTCOMES:
User Satisfaction | A user satisfaction survey will be administered at the end of one-week for participants enrolled in Step 1 of the study and at the end of four-weeks for participants enrolled in Step 2.
  A user satisfaction survey will be administered to evaluate the study participants' overall satisfaction with the app. This is a non-health outcome designed to better understand the user's perception of the app. The survey will consist of 20 statements that users will rate on a 1-7 Likert type scale (1=Disagree, 7= Agree). Satisfaction scores will be averaged and converted to percentages with higher percentages representing better user satisfaction with the app.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Potter, Ph.D., Principal Investigator — UT Health San Antonio
Locations (1):
- UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No